CLINICAL TRIAL: NCT04146298
Title: Clinical Trial Evaluating the Safety and Activity of Mutant KRAS G12V-specific TCR Transduced T Cell Therapy for Advanced Pancreatic Cancer
Brief Title: Mutant KRAS G12V-specific TCR Transduced T Cell Therapy for Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Doctor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChanghaiH-PP06
Record Dates: First submitted 2019-10-26; First posted 2019-10-31 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Pancreatic Neoplasms; Pancreatic Ductal Adenocarcinoma; Advanced Cancer
Keywords: pancreatic cancer; TCR transduced T cells; adoptive cell therapy; KRAS
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide; fludarabine; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR Transduced T cell therapy (Experimental): Pre-conditioning: Non-myeloablative, lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine
  TCR transduced T cell infusion: mutant KRAS G12V-specific TCR transduced autologous T cells (1e9~1e11). If the participant responds to the first infusion, the second or more infusions will be considered when the disease is progressing.
  Anti-PD-1 therapy: anti-PD-1 will be administered if needed.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Mutant KRAS G12V-specific TCR transduced autologous T cells; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be administered prior to cell infusion.
Drug: Fludarabine — Fludarabine will be administered prior to cell infusion.
Biological: Mutant KRAS G12V-specific TCR transduced autologous T cells — After preconditioning regimen, T cells will be infused to the patient intravenously in the Patient Care Unit over approximately 30 to 50 minutes.
Drug: Anti-PD-1 monoclonal antibody — During the treatment, anti-PD-1 monoclonal antibody will be administered if needed.
  Other Names: Anti-PD-1

SUMMARY:
This clinical trial will evaluate the safety and activity of mutant KRAS G12V-specific TCR transduced T cell therapy for advanced pancreatic cancer patients who express the KRAS G12V mutation and HLA-A*11:01 allele. The theoretical basis of this study is that mutant KRAS antigen-specific TCR transduced autologous Tcells will target and kill HLA-matched mutant KRAS cancer cells but not normal cells.

DETAILED DESCRIPTION:
Hotspot KRAS mutations exist in various cancers, especially pancreatic, lung and colorectal cancer. Mutations in KRAS are implicated in the development of pancreatic cancer and are associated with poor prognosis of the patients. KRAS is an attractive target for cancer treatment because it is a driver mutation and is likely expressed by all cells in a tumor. Recently,T cells targeting mutant KRAS have been identified in patients with epithelial cancers, and these T-cell receptors (TCR) have been characterized. For example, TCRs that target mutant KRAS G12D peptides presented by HLA-C*08:02, and a TCR that targets a KRAS G12V peptide presented by HLA-A*11:01 have been identified. Mutant KRAS-reactive T cells appear capable of inducing tumor regression as highlighted in a patient with metastatic colorectal cancer who experienced regression of metastatic tumors after infusion of HLA-C*08:02-restricted KRAS-G12D reactive tumor-infiltrating lymphocytes (TIL). The investigators will test the safety and activity of adoptive transfer of autologous T cells genetically engineered to express a TCR that targets mutant KRAS G12V in the context of HLA-A*11:01 in HLA-matched patients with advanced pancreatic cancer that express mutant KRAS G12V. The investigators will also measure the in vivo survival of engineered T cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable and pathologically confirmed advanced pancreatic cancer, including metastatic pancreatic cancer (who have received standard chemotherapy) and recurrent pancreatic cancer (who have received surgery and adjuvant chemotherapy previously).
* Patient's tumor must express the KRAS G12V mutation, or a G12V mutation in HRAS or NRAS, as determined by DNA or RNA sequencing methods.
* Patients must be HLA-A*11:01.
* Patients with brain metastasis may be eligible if they are asymptomatic and there are fewer than 3 brain lesions that are each less than 1 cm in diameter.
* Patients between 18 to 75 years old are eligible.
* Patients should have good clinical performance status (ECOG 0 or 1).
* Patients must practice birth control once enrolled into the study and for up to four months after therapy.
* Patients must be seronegative for HIV antibody.
* Patients must be seronegative for hepatitis B surface antigen and core antibody (or HBV non-detectable by QPCR).
* Patients must be seronegative for hepatitis C antibody (or HCV non-detectable by QPCR).
* Baseline hematology criteria:

  * Absolute neutrophil count of at least 1000/mm^3.
  * White blood cell count of at least 3000/mm^3.
  * Platelet count of at least 100,000/mm^3.
  * Hemoglobin > 8.0 g/dL.
* Baseline chemistry criteria:

  * Serum ALT/AST less than or equal to 3.0 x ULN.
  * Total bilirubin less than or equal to 1.5 mg/dL, unless the patient has Gilbert's Syndrome in which case total bilirubin must be less than or equal to 3.0 mg/dL.
  * Serum creatinine less than or equal to 1.6 mg/dL.
* Anticipated lifespan greater than 12 weeks.
* Patients must be willing and able to comply with all study-related procedures and follow-up requirements.
* Patients must be able to understand and sign a written Informed Consent Document as well as a durable power of attorney.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Patients with any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease or HIV).
* Patients with active systemic infections, coagulation disorders, or any other major medical illnesses.
* Patients with concurrent opportunistic infections.
* Patients on concurrent systemic steroid therapy.
* Patients with a history of severe immediate hypersensitivity reaction to any of the medicines used in this study (e.g., cyclophosphamide, fludarabine).
* Patients with active coronary ischemic symptoms.
* Patients who are receiving any other investigational agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-related adverse events | 18 months following cell infusion
  Aggregate of all adverse events, as well as their frequency and severity
Objective response rate | From the date of cell infusion to disease progression (up to 18 months after cell infusion).
  Percentage of patients who have a clinical response to treatment (objective tumor regression)

SECONDARY OUTCOMES:
The percentage of TCR transduced T cells in peripheral blood | 1, 3, 7, 14, 28, 42 and 84 days after cell infusion, then every 3 months, and up to 18 months after cell infusion.
  The percentage of TCR transduced T cells in peripheral blood will be detected with an established flow cytometric assay.
Overall survival | From date of cell infusion until the date of death from any cause, whichever came first, assessed up to 18 months after cell infusion.
  The time between cell infusion and the death of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

REFERENCES:
- [Result] Xu X, Guo S, Gu H, Cha Z, Shi X, Yin X, Wang H, Gao S, Li B, Zhu L, Jing W, Zheng K, Shao Z, Cheng P, Zheng C, Shih YP, Li Y, Qian B, Gao D, Tran E, Jin G. Identification and validation of a T cell receptor targeting KRAS G12V in HLA-A*11:01 pancreatic cancer patients. JCI Insight. 2025 Jan 23;10(2):e181873. doi: 10.1172/jci.insight.181873. PMID 39846249
- [Result] Cafri G, Yossef R, Pasetto A, Deniger DC, Lu YC, Parkhurst M, Gartner JJ, Jia L, Ray S, Ngo LT, Jafferji M, Sachs A, Prickett T, Robbins PF, Rosenberg SA. Memory T cells targeting oncogenic mutations detected in peripheral blood of epithelial cancer patients. Nat Commun. 2019 Jan 25;10(1):449. doi: 10.1038/s41467-019-08304-z. PMID 30683863
- [Result] Tran E, Robbins PF, Lu YC, Prickett TD, Gartner JJ, Jia L, Pasetto A, Zheng Z, Ray S, Groh EM, Kriley IR, Rosenberg SA. T-Cell Transfer Therapy Targeting Mutant KRAS in Cancer. N Engl J Med. 2016 Dec 8;375(23):2255-2262. doi: 10.1056/NEJMoa1609279. PMID 27959684